CLINICAL TRIAL: NCT04652804
Title: A Precision Randomized Trial to Evaluate the Impact of Tailored Hepatitis C Virus (HCV) Treatment Adherence Support on HCV Treatment Outcomes in HIV/HCV Co-infected and HCV Mono-infected People Who Inject Drugs (PWID) in India.
Brief Title: Supporting Treatment Outcomes Among PWID
Acronym: STOP-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: YR Gaitonde Centre for AIDS Research and Education (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00232125; 5R01AI145555-02 (NIH)
Record Dates: First submitted 2020-11-20; First posted 2020-12-03 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Hepatitis C; HIV Coinfection
Keywords: Patient Navigation; Treatment Adherence; People who inject drugs (PWID); Directly Observed Therapy (DOT); India
MeSH Terms: conditions — Hepatitis C; HIV Infections; Treatment Adherence and Compliance; Directly Observed Therapy

STUDY DESIGN:
Intervention Model Description: This is a 3-arm, individual-level randomized clinical trial, in which treatment assignment probabilities vary according to participants' estimated propensity for treatment failure at baseline (precision randomization). Minimal risk individuals have a higher likelihood of being allocated to lower intensity intervention and elevated risk individuals have higher likelihood of being allocated to higher intensity intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Low Intensity Intervention (Active Comparator): 4 weeks dispensation + standard adherence counseling
  Interventions: Behavioral: Low intensity HCV treatment adherence support
- Arm 2: Medium Intensity Intervention (Active Comparator): 4 weeks dispensation + support from patient navigator
  Interventions: Behavioral: Medium intensity HCV treatment adherence support
- Arm 3: High Intensity Intervention (Active Comparator): Directly Observed Therapy with flexible dispensing and support from patient navigator
  Interventions: Behavioral: High intensity HCV treatment adherence support

INTERVENTIONS:
Behavioral: Low intensity HCV treatment adherence support — A 28-day supply of medication will be dispensed to participants at entry, 4 weeks, and 8 weeks. Participants will receive standard adherence counseling at entry and every refill pickup/home or field delivery. Participants will have access to all of the services available at the ICC including facilitated linkage to referrals as needed. Site staff will routinely track clients who miss refill appointments in real-time using standard tracking measurements
  Arms: Arm 1: Low Intensity Intervention
Behavioral: Medium intensity HCV treatment adherence support — The medium intensity intervention will include standard of care dispensation of a 28-day supply of medication at entry, 4 weeks and 8 weeks. Participants will be assigned to a patient navigator (PN) and receive tailored patient navigation support for medication reminders, picking up medication refills (or home or field delivery of study medications), overcoming barriers as well as service linkage. Participant will be contacted by the PN at least once every two weeks.
  Arms: Arm 2: Medium Intensity Intervention
Behavioral: High intensity HCV treatment adherence support — The high intensity intervention will involve patient-centered DOT with flexibility in terms of the frequency of pickup and the site of DOT (ICC, field-based) with a minimum of at least 1 observed dose per week. Participants in this arm will also receive PN support for overcoming barriers and service linkage similar to participants in Arm 2. The main differences between Arms 2 and 3 are: (i) medications will not be dispensed for more than one week at a time (to coincide with opioid agonist therapy (OAT) dosing, where applicable); and (ii) ≥1 dose/week will be observed.
  Arms: Arm 3: High Intensity Intervention

SUMMARY:
The goal of this study is to improve HCV care continuum outcomes for people who inject drugs (PWID), reduce potential onward transmission to others and improve HIV outcomes among those who are HIV/HCV coinfected. The study will evaluate whether HCV treatment outcomes (sustained virologic response, treatment completion, adherence) and post treatment outcomes (HCV reinfection, HIV viral suppression) in HCV mono- and HIV/HCV co-infected PWID can be optimized by tailoring treatment support in 7 PWID-focused integrated HIV/HCV prevention and treatment centers in India.

DETAILED DESCRIPTION:
The primary objective is to evaluate whether the intensity of treatment adherence support affects sustained virologic response rates in HCV mono- and HIV/HCV co-infected participants receiving HCV direct-acting antivirals (DAA) in PWID-focused centers. Secondary objectives are: 1. To evaluate whether the intensity of treatment adherence support affects HCV treatment completion rates. 2. To evaluate whether the intensity of treatment adherence support affects HCV treatment adherence. 3. To estimate the incidence and correlates of HCV reinfection among HCV mono- and HIV/HCV coinfected PWID who achieve HCV cure. 4. To evaluate the impact of HCV cure on HIV viral suppression among HIV/HCV coinfected PWID.

Investigators will evaluate this via a 3-arm, individual-level randomized clinical trial, in which treatment assignment probabilities vary according to participants' estimated propensity for treatment failure at baseline (precision randomization). An estimated 3,000 persons will be enrolled and randomized at 7 community-based integrated care centers (ICCs) across India across a duration of 18 - 24 months. Data from these 7 ICCs on early HIV treatment refills/viral suppression (3-6 months after antiretroviral therapy (ART) initiation) will be used to develop and validate an algorithm to predict propensity for HCV treatment failure. Prior to treatment initiation, each participant will undergo a questionnaire to capture information on barriers/ facilitators to treatment adherence identified in the prediction model in order to determine the propensity for HCV treatment failure (minimal or elevated risk). Individuals will be preferentially randomized to the support level that matches their failure risk. Those at elevated risk for treatment failure will be randomized at an allocation ratio of 3:2:1 for Arm 3 (high intensity support), Arm 2 (medium intensity support) and Arm 1 (low intensity support), respectively. Conversely, those at minimal risk will be randomized at a ratio of 1:2:3 to Arm 3 (high intensity support), Arm 2 (medium intensity support) and Arm 1 (low intensity support), respectively. Participants and study staff will be blinded to the risk classification (minimal, elevated) but, because of the nature of the interventions, blinding to intervention assignment is not possible.

Persons will be treated for HCV according to the standard of care in India. Minimal laboratory monitoring will be used except when clinically indicated. Participants with decompensated cirrhosis will be excluded from treatment.

All HIV/HCV co-infected participants and those HCV monoinfected participants who achieve SVR will be followed post-treatment. These individuals will be followed every six months after the SVR assessment to assess HCV reinfection and HIV viral suppression (among HIV/HCV coinfected participants) for up to 30 months after SVR.

ELIGIBILITY:
Inclusion Criteria:

* Registered for care at an Integrated Care Center (ICC) in one of the 7 field sites.
* Active HCV infection confirmed by a detectable HCV RNA by polymerase chain reaction (PCR) (HCV RNA ≥ 30 copies/ml) within 90 days prior to study entry.
* Liver disease stage defined as non-cirrhotic or compensated cirrhotic (metric/diagnostic criteria used for fibrosis staging) within 90 days prior to study entry.

  i. Albumin >3.0 g/L. ii. Hemoglobin >8.0 g/dL for women; >9.0 g/dL for men. iii. Platelet count >50,000/mm3. iv. Calculated creatinine clearance (CrCl) using Cockcroft-Gault method >30 mL/min. v. Aspartate aminotransferase (AST/SGOT) <10 times the upper limit of the normal range (ULN). vi. Alanine aminotransferase (ALT/SGPT) <10 times the ULN. vii. Total bilirubin <1.5 times the ULN for participants not on atazanavir (ATV) and <3 times the ULN for participants on ATV. viii. International normalized ratio (INR) <1.5 times the ULN.
* Life expectancy greater than 1 year (as determined by study clinician)
* Willing to initiate HCV treatment
* Agree to be randomized to an adherence support strategy
* Ability and willingness to provide written informed consent
* Female participants of reproductive potential must not be pregnant
* All female participants of reproductive potential must agree not to participate in a conception process
* All female participants of reproductive potential must agree to use at least one reliable form of contraceptive while receiving protocol-specified medication, and for 6 weeks after stopping the medication.

Exclusion Criteria:

* Psychologically unfit to provide written informed consent.
* Planning to migrate within the next six months.
* Known allergy/sensitivity or any hypersensitivity to components of study drug(s) or their formulation.
* Acute or serious illness requiring systemic treatment and/or hospitalization within 30 days prior to study entry.
* In HIV positive participants, presence of active or acute AIDS-defining opportunistic infections within 30 days prior to study entry.
* Use of prohibited medications within the past 14 days prior to study entry.
* Evidence of decompensated liver disease on clinical exam.
* Evidence of active tuberculosis.
* Evidence of chronic hepatitis B infection (HBsAg positive).
* Currently on HCV treatment.
* Prior history of DAA-based HCV treatment
* Confirmed active SARS CoV-2 infection or suspected active SARS CoV-2 infection at enrollment.
* Currently nursing (breastfeeding).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil S Solomon, PhD MBBS MPH, Principal Investigator — Johns Hopkins University School of Medicine and Y.R. Gaitonde Centre for AIDS Research and Education; Shruti H Mehta, PhD MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- YR Gaitonde Centre for AIDS Research and Education, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehta SH, Lau BM, Ehrhardt S, McFall A, Gunaratne MP, Baishya J, Kedar A, Srikrishnan AK, Evans J, Loeb T, Pradeep A, Kumar MS, Thomas DL, Lucas GM, Solomon SS. A precision randomized trial to evaluate the impact of tailored hepatitis C treatment adherence support on HCV treatment outcomes among people who inject drugs in India: design and baseline characteristics of the STOP-C trial. Am J Epidemiol. 2025 Oct 7;194(10):2986-2998. doi: 10.1093/aje/kwae430. PMID 39572371

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Low Intensity Intervention (Minimal Risk): 4 weeks dispensation + standard adherence counseling
  Low intensity Hepatitis C Virus (HCV) treatment adherence support: A 28-day supply of medication will be dispensed to participants at entry, 4 weeks, and 8 weeks. Participants will receive standard adherence counseling at entry and every refill pickup/home or field delivery. Participants will have access to all of the services available at the ICC including facilitated linkage to referrals as needed. Site staff will routinely track clients who miss refill appointments in real-time using standard tracking measurements
- Arm 2: Medium Intensity Intervention (Minimal Risk); Arm 2: Medium Intensity Intervention (Elevated Risk): 4 weeks dispensation + support from patient navigator
  Medium intensity HCV treatment adherence support: The medium intensity intervention will include standard of care dispensation of a 28-day supply of medication at entry, 4 weeks and 8 weeks. Participants will be assigned to a patient navigator (PN) and receive tailored patient navigation support for medication reminders, picking up medication refills (or home or field delivery of study medications), overcoming barriers as well as service linkage. Participant will be contacted by the PN at least once every two weeks.
- Arm 3: High Intensity Intervention (Minimal Risk): Directly Observed Therapy (DOT) with flexible dispensing and support from patient navigator
  High intensity HCV treatment adherence support: The high intensity intervention will involve patient-centered DOT with flexibility in terms of the frequency of pickup and the site of DOT (ICC, field-based) with a minimum of at least 1 observed dose per week. Participants in this arm will also receive PN support for overcoming barriers and service linkage similar to participants in Arm 2. The main differences between Arms 2 and 3 are: (i) medications will not be dispensed for more than one week at a time (to coincide with opioid agonist therapy (OAT) dosing, where applicable); and (ii) ≥1 dose/week will be observed.
- Arm 1: Low Intensity Intervention (Elevated Risk): 4 weeks dispensation + standard adherence counseling
  Low intensity HCV treatment adherence support: A 28-day supply of medication will be dispensed to participants at entry, 4 weeks, and 8 weeks. Participants will receive standard adherence counseling at entry and every refill pickup/home or field delivery. Participants will have access to all of the services available at the ICC including facilitated linkage to referrals as needed. Site staff will routinely track clients who miss refill appointments in real-time using standard tracking measurements
- Arm 3: High Intensity Intervention (Elevated Risk): Directly Observed Therapy with flexible dispensing and support from patient navigator
  High intensity HCV treatment adherence support: The high intensity intervention will involve patient-centered DOT with flexibility in terms of the frequency of pickup and the site of DOT (ICC, field-based) with a minimum of at least 1 observed dose per week. Participants in this arm will also receive PN support for overcoming barriers and service linkage similar to participants in Arm 2. The main differences between Arms 2 and 3 are: (i) medications will not be dispensed for more than one week at a time (to coincide with opioid agonist therapy (OAT) dosing, where applicable); and (ii) ≥1 dose/week will be observed.
Period: Overall Study
Arm/Group | Arm 1: Low Intensity Intervention (Minimal Risk) | Arm 2: Medium Intensity Intervention (Minimal Risk) | Arm 3: High Intensity Intervention (Minimal Risk) | Arm 1: Low Intensity Intervention (Elevated Risk) | Arm 2: Medium Intensity Intervention (Elevated Risk) | Arm 3: High Intensity Intervention (Elevated Risk)
Started | 1022 | 684 | 342 | 157 | 320 | 475
Completed | 1019 | 684 | 341 | 157 | 319 | 474
Not Completed | 3 | 0 | 1 | 0 | 1 | 1
Not completed — Ineligible post randomization | 1 | 0 | 1 | 0 | 1 | 1
Not completed — Missing SVR lab results | 2 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data are stratified by risk stratum and arm. 2048 participants were assigned to the minimal risk stratum, and 952 were assigned to the elevated risk stratum.
Groups:
- Arm 1: Low Intensity Intervention (Minimal Risk); Arm 1: Low Intensity Intervention (Elevated Risk): 4 weeks dispensation + standard adherence counseling
  Low intensity HCV treatment adherence support: A 28-day supply of medication will be dispensed to participants at entry, 4 weeks, and 8 weeks. Participants will receive standard adherence counseling at entry and every refill pickup/home or field delivery. Participants will have access to all of the services available at the ICC including facilitated linkage to referrals as needed. Site staff will routinely track clients who miss refill appointments in real-time using standard tracking measurements
- Arm 3: High Intensity Intervention (Minimal Risk); Arm 3: High Intensity Intervention (Elevated Risk): Directly Observed Therapy with flexible dispensing and support from patient navigator
  High intensity HCV treatment adherence support: The high intensity intervention will involve patient-centered DOT with flexibility in terms of the frequency of pickup and the site of DOT (ICC, field-based) with a minimum of at least 1 observed dose per week. Participants in this arm will also receive PN support for overcoming barriers and service linkage similar to participants in Arm 2. The main differences between Arms 2 and 3 are: (i) medications will not be dispensed for more than one week at a time (to coincide with opioid agonist therapy (OAT) dosing, where applicable); and (ii) ≥1 dose/week will be observed.
- Total: Total of all reporting groups
Arm/Group | Arm 1: Low Intensity Intervention (Minimal Risk) | Arm 2: Medium Intensity Intervention (Minimal Risk) | Arm 3: High Intensity Intervention (Minimal Risk) | Arm 1: Low Intensity Intervention (Elevated Risk) | Arm 2: Medium Intensity Intervention (Elevated Risk) | Arm 3: High Intensity Intervention (Elevated Risk) | Total
Number analyzed (Participants) | 1019 | 684 | 341 | 157 | 319 | 474 | 2994
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Median (Inter-Quartile Range)
  years | 31 [26 to 36] | 30 [25 to 35] | 32 [25 to 37] | 28 [24 to 31] | 27 [23 to 30] | 27 [23 to 30] | 29 [25 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 14 | 7 | 0 | 0 | 0 | 42
  Male | 998 | 670 | 334 | 157 | 319 | 474 | 2952
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1019 | 684 | 341 | 157 | 319 | 474 | 2994
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Living with HIV [Count of Participants; unit: Participants] | 166 | 136 | 54 | 48 | 94 | 143 | 641
HCV viral load [Median (Inter-Quartile Range); unit: IU/ml] | 271186 [44108 to 724679] | 336331 [56894 to 806405] | 250493 [46659 to 734095] | 230803 [35653 to 615107] | 413023 [74639 to 921452] | 220090 [37862 to 691424] | 286574 [48859 to 769198]

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virologic Response (SVR) by Intervention Group Stratified by Defined Risk for Treatment Failure (Minimal vs Elevated)
Description: The percentage of participants who achieved SVR defined as HCV RNA < lower limit of quantification (LLOQ). HCV RNA < lower limit of quantification (LLOQ, 30 IU/ml) was measured 12 weeks (range 10 - 60 weeks) after treatment completion.
Time Frame: Between 10 and 60 weeks after scheduled end of treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1 : Low Intensity Intervention (Elevated Risk): 4 weeks dispensation + standard adherence counseling
  Low intensity HCV treatment adherence support: A 28-day supply of medication will be dispensed to participants at entry, 4 weeks, and 8 weeks. Participants will receive standard adherence counseling at entry and every refill pickup/home or field delivery. Participants will have access to all of the services available at the ICC including facilitated linkage to referrals as needed. Site staff will routinely track clients who miss refill appointments in real-time using standard tracking measurements
- Arm 2: Medium Intervention (Elevated Risk): 4 weeks dispensation + support from patient navigator
  Medium intensity HCV treatment adherence support: The medium intensity intervention will include standard of care dispensation of a 28-day supply of medication at entry, 4 weeks and 8 weeks. Participants will be assigned to a patient navigator (PN) and receive tailored patient navigation support for medication reminders, picking up medication refills (or home or field delivery of study medications), overcoming barriers as well as service linkage. Participant will be contacted by the PN at least once every two weeks.
Arm/Group | Arm 1: Low Intensity Intervention (Minimal Risk) | Arm 2: Medium Intensity Intervention (Minimal Risk) | Arm 3: High Intensity Intervention (Minimal Risk) | Arm 1 : Low Intensity Intervention (Elevated Risk) | Arm 2: Medium Intervention (Elevated Risk) | Arm 3: High Intensity Intervention (Elevated Risk)
Number analyzed (Participants) | 1019 | 684 | 341 | 157 | 319 | 474
Participants | 638 | 416 | 233 | 76 | 145 | 241
Statistical Analysis 1: Comparison: Arm 1: Low Intensity Intervention (Minimal Risk) vs Arm 3: High Intensity Intervention (Minimal Risk); Reference group: Low Intensity Intervention; Test type: Superiority; Risk Ratio (RR) = 1.09, 95% CI 2-sided [1.00 to 1.19]
Statistical Analysis 2: Comparison: Arm 1: Low Intensity Intervention (Minimal Risk) vs Arm 2: Medium Intensity Intervention (Minimal Risk); Reference Group: Low Intensity Intervention; Test type: Superiority; Risk Ratio (RR) = 0.97, 95% CI 2-sided [0.90 to 1.05]
Statistical Analysis 3: Comparison: Arm 1 : Low Intensity Intervention (Elevated Risk) vs Arm 3: High Intensity Intervention (Elevated Risk); Reference group: High Intensity Intervention; Test type: Superiority; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.80 to 1.15]
Statistical Analysis 4: Comparison: Arm 2: Medium Intervention (Elevated Risk) vs Arm 3: High Intensity Intervention (Elevated Risk); Reference group: High Intensity Intervention; Test type: Superiority; Risk Ratio (RR) = 0.89, 95% CI 2-sided [0.77 to 1.04]

2. Secondary Outcome: HCV Treatment Completion
Description: The percentage of participants who completed the prescribed course of treatment (12 or 24 weeks). Participants with compensated cirrhosis and genotype 3 infection would have received 24 weeks of treatment. All other participants would have received treatment for 12 weeks. All participants in this study received 12 weeks of treatment.
Time Frame: Measured at the end of prescribed course of treatment (12 or 24 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Low Intensity Intervention (Minimal Risk) | Arm 2: Medium Intensity Intervention (Minimal Risk) | Arm 3: High Intensity Intervention (Minimal Risk) | Arm 1 : Low Intensity Intervention (Elevated Risk) | Arm 2: Medium Intervention (Elevated Risk) | Arm 3: High Intensity Intervention (Elevated Risk)
Number analyzed (Participants) | 1019 | 684 | 341 | 157 | 319 | 474
Participants | 969 | 660 | 311 | 138 | 291 | 413

3. Secondary Outcome: Adherence >90% (Self-report)
Description: The percentage of participants who self-report taking >90% of doses during treatment.
Time Frame: Measured at the end of prescribed course of treatment (12 or 24 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Low Intensity Intervention (Minimal Risk) | Arm 2: Medium Intensity Intervention (Minimal Risk) | Arm 3: High Intensity Intervention (Minimal Risk) | Arm 1 : Low Intensity Intervention (Elevated Risk) | Arm 2: Medium Intervention (Elevated Risk) | Arm 3: High Intensity Intervention (Elevated Risk)
Number analyzed (Participants) | 1019 | 684 | 341 | 157 | 319 | 474
Participants | 860 | 595 | 284 | 105 | 239 | 372

4. Secondary Outcome: Adherence >90% (Medication Records)
Description: The percentage of participants in possession of >90% of doses during treatment based on medication refills and pill counts.
Time Frame: Measured at the end of prescribed course of treatment (12 or 24 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Low Intensity Intervention (Minimal Risk) | Arm 2: Medium Intensity Intervention (Minimal Risk) | Arm 3: High Intensity Intervention (Minimal Risk) | Arm 1 : Low Intensity Intervention (Elevated Risk) | Arm 2: Medium Intervention (Elevated Risk) | Arm 3: High Intensity Intervention (Elevated Risk)
Number analyzed (Participants) | 1019 | 684 | 341 | 157 | 319 | 474
Participants | 755 | 541 | 234 | 99 | 233 | 305

5. Secondary Outcome: Adherence Level (Self-report)
Description: The percentage of doses taken during treatment as self-reported by the participant.
Time Frame: Measured at the end of prescribed course of treatment (12 or 24 weeks)
Measure: Median (Inter-Quartile Range); unit: % of doses taken
Arm/Group | Arm 1: Low Intensity Intervention (Minimal Risk) | Arm 2: Medium Intensity Intervention (Minimal Risk) | Arm 3: High Intensity Intervention (Minimal Risk) | Arm 1 : Low Intensity Intervention (Elevated Risk) | Arm 2: Medium Intervention (Elevated Risk) | Arm 3: High Intensity Intervention (Elevated Risk)
Number analyzed (Participants) | 1019 | 684 | 341 | 157 | 319 | 474
% of doses taken | 100 [98.7 to 100] | 100 [100 to 100] | 100 [100 to 100] | 100 [83.3 to 100] | 100 [90.0 to 100] | 100 [93.3 to 100]

6. Secondary Outcome: Adherence Level (Medication Records)
Description: The percentage of doses participants had in their possession during treatment based on medication refills and pill counts.
Time Frame: Measured at the end of prescribed course of treatment (12 or 24 weeks)
Measure: Median (Inter-Quartile Range); unit: Percentage of doses
Arm/Group | Arm 1: Low Intensity Intervention (Minimal Risk) | Arm 2: Medium Intensity Intervention (Minimal Risk) | Arm 3: High Intensity Intervention (Minimal Risk) | Arm 1 : Low Intensity Intervention (Elevated Risk) | Arm 2: Medium Intervention (Elevated Risk) | Arm 3: High Intensity Intervention (Elevated Risk)
Number analyzed (Participants) | 1019 | 684 | 341 | 157 | 319 | 474
Percentage of doses | 96.5 [89.4 to 98.8] | 96.6 [91.3 to 98.8] | 95.2 [87.4 to 98.8] | 93.3 [85.6 to 97.6] | 95.5 [89.2 to 98.8] | 92.9 [84.9 to 97.6]

7. Secondary Outcome: HCV Reinfection
Description: The percentage of participants who test positive for HCV Core Antigen after achieving SVR.
Time Frame: Measured at 6 month intervals after confirmation of SVR for up to 36 months.
Reporting Status: Not Posted

8. Secondary Outcome: HIV Viral Suppression Among HIV/HCV Coinfected Participants
Description: The percentage of HIV/HCV co-infected participants with HIV RNA less than LLOQ after the SVR assessment. HCV RNA abstracted from chart reviews.
Time Frame: After assessment of SVR for up to 36 months.
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Exploratory Outcome Measure: Medication for Opioid Use Disorder (MOUD) Initiation
Description: Rate of MOUD Initiation post randomization
Time Frame: Measured daily from Entry Visit to post SVR for up to 36 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Exploratory Outcome Measure: Medication for Opioid Use Disorder Retention
Description: Consistent MOUD use post randomization
Time Frame: Measured daily from Entry Visit to post SVR for up to 36 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Exploratory Outcome Measure: Quality of Life
Description: Self-reported quality of life score based on self-report
Time Frame: Measured at 6 month intervals at the SVR visit and post SVR for up to 36 months.
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Exploratory Outcome Measure: Mortality
Description: Mortality rate per person years
Time Frame: Measured from Entry visit to post SVR for up to 36 months.
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Exploratory Outcome Measure: Cost Effectiveness of Tailored Support Options (Low, Medium and High Intensity)
Description: Incremental cost effectiveness ratios calculated between an intervention and its next least costly comparator and assessed against per capita Gross Domestic Product (GDP)
Time Frame: Measured at weekly intervals starting from Entry visit to SVR visit (up to 12 weeks after treatment completion).
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Exploratory Outcome Measure: Acceptability of Low, Medium and High Intensity Interventions
Description: Measured by in-depth qualitative interviews with integrated care clinic staff and clients post intervention.
Time Frame: Qualitative interviews will be conducted between the end of treatment visit and the SVR visit (up to 12 weeks after treatment completion).
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From date of randomization up to the expected Sustained Virologic Response (SVR) 12 week visit date
Description: All AEs that occurred after the entry visit and up to SVR evaluation were recorded if any of the following criteria were met:
  * All grade ≥ 3 AEs
  * All AEs that led to a change in treatment/intervention regardless of grade
  * All AEs meeting SAE definition or expedited adverse event (EAE) reporting requirement All AEs that were reported had their severity graded as per Division of AIDS guidelines. Serious adverse events (SAE) was reported within 7 days of when the site staff were notified.
Arm/Group | Arm 1: Low Intensity Intervention (Minimal Risk) | Arm 2: Medium Intensity Intervention (Minimal Risk) | Arm 3: High Intensity Intervention (Minimal Risk) | Arm 1: Low Intensity Intervention (Elevated Risk) | Arm 2: Medium Intensity Intervention (Elevated Risk) | Arm 3: High Intensity Intervention (Elevated Risk)
All-Cause Mortality (participants affected / at risk) | 9/1022 | 3/684 | 3/342 | 4/157 | 9/320 | 7/475
Serious Adverse Events (participants affected / at risk) | 14/1022 | 5/684 | 4/342 | 7/157 | 10/320 | 11/475
Other Adverse Events (participants affected / at risk) | 1/1022 | 1/684 | 2/342 | 1/157 | 0/320 | 1/475
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Low Intensity Intervention (Minimal Risk) (N=1022) | Arm 2: Medium Intensity Intervention (Minimal Risk) (N=684) | Arm 3: High Intensity Intervention (Minimal Risk) (N=342) | Arm 1: Low Intensity Intervention (Elevated Risk) (N=157) | Arm 2: Medium Intensity Intervention (Elevated Risk) (N=320) | Arm 3: High Intensity Intervention (Elevated Risk) (N=475)
Death (General disorders) | 9 (9) | 3 (3) | 3 (3) | 4 (4) | 9 (9) | 7 (7)
Event other than death (General disorders) | 5 (5) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Low Intensity Intervention (Minimal Risk) (N=1022) | Arm 2: Medium Intensity Intervention (Minimal Risk) (N=684) | Arm 3: High Intensity Intervention (Minimal Risk) (N=342) | Arm 1: Low Intensity Intervention (Elevated Risk) (N=157) | Arm 2: Medium Intensity Intervention (Elevated Risk) (N=320) | Arm 3: High Intensity Intervention (Elevated Risk) (N=475)
Event other than death (General disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT04652804/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT04652804/SAP_001.pdf